CLINICAL TRIAL: NCT02043483
Title: Obstructive Sleep Apnoea and Associated Metabolic/Cardiovascular Disorders: Understanding Mechanisms Towards Early Diagnosis and Prognosis
Brief Title: Identification of Biomarkers for Obstructive Sleep Apnoea Syndrome
Status: Completed | Type: Observational
Sponsor: Universidade Nova de Lisboa (Other)
Collaborators: Centro de Estudos de Doenças Crónicas (Other); NOVA Medical School (Other); Centro Hospitalar Lisboa Norte (Other); Instituto Nacional de Saúde Dr. Ricardo Jorge (Unknown); Biotempo (Unknown); Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Other Study IDs: FCM-
Record Dates: First submitted 2013-11-12; First posted 2014-01-23 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Obstructive Sleep Apnoea Syndrome
Keywords: CPAP; OSAS; CEDOC (Centro de Estudos de Doenças Crónicas); FCM (Faculdade de Ciências Médicas); UNL (Universidade Nova de Lisboa; NOVA MEDICAL SCHOOL; FCT (Fundação para a Ciência e Tecnologia)
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- CPAP: Patients with moderate/severe OSAS will be treated with CPAP
- Control: Patients with snoring will not be subject to treatment with CPAP

SUMMARY:
Untreated Obstructive Sleep Apnea Syndrome (OSAS) has long-term complications, namely metabolic imbalances (obesity, dislipidemia, type 2 diabetes mellitus). Until now, no molecular markers for this physiopathological connection have been identified.

This project aims to determine non-invasive biomarkers that may allow better comprehension of the metabolic consequences of OSAS, as well as assess the effect of Continuous positive airway pressure (CPAP) on these metabolic parameters.

This project will integrate the clinical, metabolic, genetic/proteomic and biologic systems to further explore the mechanisms behind OSAS, as well as the effect of the treatment with CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Male
* 25-60 years
* Mild/Moderate/Severe OSAS

Exclusion Criteria:

* Female
* Other sleep disorders
* Previous CPAP therapy
* Type 1 diabetes mellitus
* Familiar Dyslipidemia
* Severe organ pathology
* Acute disease

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Obstructive Sleep Apnoea Syndrome Males 25-60 years
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with clinical improvement | 6 months
  Treatment efficacy of CPAP will be assessed at the end of treatment through a clinical observation.

SECONDARY OUTCOMES:
Frequency of occurence of biomarkers | 6 months
  Using Mass Spectrometric Immunoassay, we will identify which biomarkers have a positive association with long-term treatment effect.

CONTACTS AND LOCATIONS:
Overall Officials: Amélia Feliciano, MD, Principal Investigator — Centro Hospitalar Lisboa Norte
Locations (1):
- Centro Hospitalar Lisboa Norte, Lisbon, Portugal